CLINICAL TRIAL: NCT02235402
Title: A Randomised, Parallel-group, Double-blind, Double-dummy Study to Compare the Effects of Lacidipine Versus Bendrofluazide on Markers of Platelet Activation and Haemorheological Factors in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231.336
Record Dates: First submitted 2014-09-09; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — lacidipine; Bendroflumethiazide

ARMS (3):
- Lacidipine (Experimental)
  Interventions: Drug: Lacidipine
- Bendrofluazide (Active Comparator)
  Interventions: Drug: Bendrofluazide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lacidipine
  Arms: Lacidipine
Drug: Bendrofluazide
  Arms: Bendrofluazide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to compare the effects of lacidipine on markers of platelet activation and other rheological factors in hypertensive patients with those of bendrofluazide

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Hypertensive at screening: Diastolic blood pressure (DBP) 95 - 115 mm Hg and / or systolic blood pressure (SBP) >= 160 mm Hg on no therapy or on monotherapy. If currently on monotherapy, DBP could have been < 95 mm Hg and SBP < 160 mm Hg, but the patient must have been experiencing unacceptable side effects from their current treatment. Patient must then be able to stop treatment for the placebo run in phase of four weeks without endangering their health (at investigator's discretion)
* Hypertensive at randomisation: DBP 95-115 mm Hg and or SBP >=160
* Able to give written informed consent

Exclusion Criteria:

* Grad III or grad IV hypertensive retinopathy
* Renal impairment; serum creatinine > 150 µmol/L
* Heart failure. (New York Heart Association (NYHA) Class III or IV)
* Liver impairment (abnormal Liver function test (LFT) with aspartate-amino transferase (AST) / alanine-amino transferase (ALT) > 2x upper normal limit or bilirubin > 2x upper normal limit)
* Recent (< 2 months) history of unstable angina
* Recent (< 2 months) history of myocardial infarction
* Recent (< 2 months) history of stroke
* History of diabetes mellitus or impaired glucose tolerance or random blood glucose >= 9 mMol/L
* Any acute systemic illness or infection
* Any severe disease which could interfere with survival or well-being during the study (e.g. malignancy)
* Patients of child bearing potential
* Current or previous drug and / or alcohol abuse
* Severely limited venous access
* Haemoglobin < 10g/dL (male patients), haemoglobin < 9g/dL (female patients)
* Requirement for anticoagulant therapy
* Severe valvular heart disease (investigator's discretion)
* Atrial fibrillation or other serious cardiac dysrhythmia
* History of thyroid disease or abnormal thyroid function test (thyroid stimulating hormone (TSH) < 0.4 mU/L or > 5.4 mU/L)
* History of connective tissue disorder
* Concurrent participation in any other clinical trial or participation within two months enrolment
* Requirement for restricted drugs
* Patients currently on treatment with lacidipine or bendrofluazide (BNFZ)
* Patients unable to attend clinics
* Any clinical condition which in the opinion of the investigator, would preclude the safe fulfillment of the protocol and the safe administration of trial medication
* Seated blood pressure (BP) exceeding either 210 mm Hg (systolic) or 115 mm Hg (diastolic) at screening or randomization
* Standing BP < 140 mm Hg (systolic) and < 95 mm Hg (diastolic) at randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1997-12; Primary Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Changes in ß-TG (thromboglobulin) | Up to week 12 after drug administration

SECONDARY OUTCOMES:
Changes in soluble p-selectin | Up to week 12 after drug administration
Changes in rheological factors | Up to week 12 after drug administration
Changes in lipid levels between randomisation and last visit | Up to week 12 after drug administration
Number of patients with clinical significant findings in laboratory parameters | Up to week 12 after drug administration
Number of patients with adverse events | Up to week 12 after drug administration